CLINICAL TRIAL: NCT04053699
Title: A Prospective, Multicenter, Non-Interventional Study Evaluating the Bleeding Incidence in Patients With Von Willebrand Disease Undergoing On-Demand Treatment
Brief Title: Bleeding Incidence in VWD Patients Undergoing On-Demand Treatment
Status: Completed | Type: Observational
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Other Study IDs: WIL-29
Record Dates: First submitted 2019-07-23; First posted 2019-08-12 (Actual); Results first posted 2023-12-07 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-03

CONDITIONS: Von Willebrand Diseases
MeSH Terms: conditions — von Willebrand Diseases | interventions — von Willebrand Factor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing treatment with a VWF-containing product: Patients with type 3, type 2 (except 2N), or severe type 1 VWD undergoing routine on-demand treatment with a VWF-containing product over a period of 6 months
  Interventions: Drug: Von Willebrand Factor-Containing Product

INTERVENTIONS:
Drug: Von Willebrand Factor-Containing Product — Active substances: VWF concentrates, VWF/FVIII concentrates, Cryoprecipitate VWF-containing products licensed in each participating country

SUMMARY:
The purpose of this study is to prospectively obtain reliable data on the bleeding and treatment pattern of patients with VWD undergoing on-demand treatment with a VWF-containing product over a period of 6 months. The data obtained will be used as a basis for historical comparisons with the bleeding and treatment pattern obtained from a clinical study on the efficacy of prophylactic treatment with a VWF/FVIII concentrate.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet all of the following criteria are eligible for the study:

* Male or female patients aged ≥5.5 years at the time of enrolment
* VWD type 1 (baseline von Willebrand factor activity [VWF:RCo], <30 IU/dL), 2A, 2B, 2M, or 3 according to medical history requiring substitution therapy with a VWF-containing product to control bleeding
* Currently receiving frequent on-demand treatment with a VWF-containing product
* In female patients of child-bearing potential using hormonal contraception, the medication class should remain unchanged for the duration of their study participation
* Voluntarily given, fully informed written and signed consent obtained before collection of any patient data

Exclusion Criteria:

Patients who meet any of the following criteria are not eligible for the study:

* Patients currently on prophylaxis for VWD (except for perioperative prophylaxis) as well as patients having received treatment once a month for menstrual bleeding, but not for any other bleeds
* Patients whose VWD treatment is planned to be switched from on-demand to prophylactic treatment in the next 6 months
* History, or current suspicion, of VWF or FVIII inhibitors
* Medical history of a thromboembolic event within 6 months before enrolment
* Severe liver or kidney diseases as described in the medical records
* Female patients with an existing or suspected pregnancy or who are breast-feeding at the time of enrolment
* Change in hormonal contraception within 6 months before enrolment
* Cervical or uterine conditions causing abnormal uterine bleeding (including infection or dysplasia)
* Other coagulation disorders or bleeding disorders due to anatomical reasons
* Participation in an interventional clinical study during the 6-month of study period
* Inability to complete the patient diary to reliably evaluate the type, frequency, and treatment of BEs during the 6-month study period

Min Age: 66 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Overall, 55 previously treated patients aged ≥5.5 years at the time of enrolment, with type 3, type 2 (except 2N), or severe type 1 VWD will be included into this study. Of these 55 patients, at least 6 should have type 3 VWD and at least 6 should be ≥5.5 to <16 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Solomon, MD, Study Director — Octapharma
Locations (15):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States
- Republican Research Center for Radiation Medicine and Human Ecology, Homyel, Belarus
- Bulgaria (2):
  - Specialized Hospital for Active Treatment of Haematological Diseases" EAD, Sofia, Sofia
  - "UMHAT Sveta Marina" EAD., Varna
- University Hospital Centre Zagreb, Zagreb, Croatia
- Hungary (3):
  - Medical Centre Hungarian Defence Forces, Budapest
  - Debreceni Egyetem Klinikai Központ, Regionális Haemophilia és Thrombophilia Központ, Debrecen
  - University Clinical Center, Department of Internal Medicine, Hematology, Pécs
- Lebanon (3):
  - Hotel Dieu de France Hospital, Beirut
  - American University of Beirut Medical Center, Beirut
  - Nini Hospital, Tripoli
- Russia (2):
  - Federal State Budgetary Scientific Institution Kirov Scientific-Research Institute of Hematology and Blood Transfusion of Federal, Kirov
  - Morosovskaya Children Clinical Hospital, Moscow Health Department, Department of General Hematology with the Pathology of Hemostasis, Moscow
- Ukraine (2):
  - State Institution "National Children's Specialized Hospital "OKHMATDYT" of the Ministry of Health of Ukraine," Center of Hemostasis Pathology, Kyiv
  - Community Institution of Lviv Oblast Council "West-Ukrainian Specialized Children's Medical Center, Lviv

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sadler JE. A revised classification of von Willebrand disease. For the Subcommittee on von Willebrand Factor of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Thromb Haemost. 1994 Apr;71(4):520-5. PMID 8052974
- [Background] Rodeghiero F, Castaman G, Tosetto A. How I treat von Willebrand disease. Blood. 2009 Aug 6;114(6):1158-65. doi: 10.1182/blood-2009-01-153296. Epub 2009 May 27. PMID 19474451
- [Background] Castaman G, Goodeve A, Eikenboom J; European Group on von Willebrand Disease. Principles of care for the diagnosis and treatment of von Willebrand disease. Haematologica. 2013 May;98(5):667-74. doi: 10.3324/haematol.2012.077263. PMID 23633542
- [Background] Mondorf W, Siegmund B, Mahnel R, Richter H, Westfeld M, Galler A, Pollmann H. Haemoassist--a hand-held electronic patient diary for haemophilia home care. Haemophilia. 2009 Mar;15(2):464-72. doi: 10.1111/j.1365-2516.2008.01941.x. Epub 2009 Feb 16. PMID 19226411
- [Background] Broderick CR, Herbert RD, Latimer J, Mathieu E, van Doorn N, Curtin JA. Feasibility of short message service to document bleeding episodes in children with haemophilia. Haemophilia. 2012 Nov;18(6):906-10. doi: 10.1111/j.1365-2516.2012.02869.x. Epub 2012 Jun 11. PMID 22681182
- [Background] Sholapur NS, Barty R, Wang G, Almonte T, Heddle NM. A survey of patients with haemophilia to understand how they track product used at home. Haemophilia. 2013 Sep;19(5):e289-95. doi: 10.1111/hae.12170. Epub 2013 May 15. PMID 23672744
- [Background] Maruish M. User's manual for the SF-36v2 Health Survey (3rd edition). Optum Incorporated; 2011.
- [Background] Saris-Baglama, R,DeRosa, M, Raczek, A, Bjorner, J,Turner-Bowker, D, Ware, J. The SF-10™ Health Survey for Children: A User's Guide. QualityMetric Incorporated; 2007.
- [Background] Hays RD, Spritzer KL, Schalet BD, Cella D. PROMIS(R)-29 v2.0 profile physical and mental health summary scores. Qual Life Res. 2018 Jul;27(7):1885-1891. doi: 10.1007/s11136-018-1842-3. Epub 2018 Mar 22. PMID 29569016
- [Derived] Sidonio RF Jr, Boban A, Dubey L, Inati A, Kiss C, Boda Z, Lissitchkov T, Nemes L, Novik D, Peteva E, Taher AT, Timofeeva MA, Vilchevska KV, Vdovin V, Werner S, Knaub S, Djambas Khayat C. von Willebrand factor/factor VIII concentrate (Wilate) prophylaxis in children and adults with von Willebrand disease. Blood Adv. 2024 Mar 26;8(6):1405-1414. doi: 10.1182/bloodadvances.2023011742. PMID 38237075

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients Undergoing On-demand Treatment With a VWF-containing Product: Patients with type 3, type 2 (except 2N), or severe type 1 Von Willebrand Disease (VWD) undergoing routine on-demand treatment with a VWF-containing product over a period of 6 months
  VWF-containing products: Active substances: VWF concentrates, VWF/FVIII concentrates, Cryoprecipitate VWF-containing products licensed in each participating country
  Fifty-six patient were screened and enrolled at 15 centers in 8 countries.
  14 patients were excluded from the efficacy analyses due to major deviations, resulting in 42 patients in the per protocol (PP) set.
Period: Full Analysis Set
Arm/Group | Patients Undergoing On-demand Treatment With a VWF-containing Product
Started | 56
Completed | 51
Not Completed | 5
Period: Per Protocol Set
Arm/Group | Patients Undergoing On-demand Treatment With a VWF-containing Product
Started | 42
Completed | 42
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Patients Undergoing On-demand Treatment With a VWF-containing Product: Patients with type 3, type 2 (except 2N), or severe type 1 VWD undergoing routine on-demand treatment with a VWF-containing product over a period of 6 months
  VWF-containing products: Active substances: VWF concentrates, VWF/FVIII concentrates, Cryoprecipitate VWF-containing products licensed in each participating country
Arm/Group | Patients Undergoing On-demand Treatment With a VWF-containing Product
Number analyzed (Participants) | 56
Age, Customized [Count of Participants; unit: Participants]
  6-11 years | 15
  12-16 years | 16
  >16 years | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 55
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Total Annualized Bleeding Rate (TABR)
Description: The total annualized bleeding rate (TABR) will be calculated as the total number of spontaneous bleeds, traumatic BEs, and other BEs occurring in the time period between the start of data collection for each patient and the Study Completion Visit, divided by the duration (in years) between the start of data collection and the Study Completion Visit. Surgery periods, and BEs occurring within these surgery periods, will be excluded from the calculation of TABR.
Time Frame: Screening through study completion (6 months)
Measure: Mean (Standard Deviation); unit: Bleeding events per year
Groups:
- Patients Undergoing On-demand Treatment With a VWF-containing Product: Patients with type 3, type 2 (except 2N), or severe type 1 VWF activity undergoing routine on-demand treatment with a VWF-containing product over a period of 6 months
  VWF-containing products: Active substances: VWF concentrates, VWF/FVIII concentrates, Cryoprecipitate VWF-containing products licensed in each participating country
Arm/Group | Patients Undergoing On-demand Treatment With a VWF-containing Product
Number analyzed (Participants) | 42
Bleeding events per year | 29.13 (22.925)

2. Secondary Outcome: Spontaneous Annualized Bleeding Rate (SABR)
Description: Spontaneous annualized bleeding rate (SABR), calculated in analogy with TABR. This includes all bleeding episodes that occurred spontaneously.
Time Frame: Screening through study completion (6 months)
Measure: Mean (Standard Deviation); unit: Bleeding events per year
Groups:
- Patients Undergoing On-demand Treatment With a VWF-containing Product: Patients with type 3, type 2 (except 2N), or severe type 1 VWD undergoing routine on-demand treatment with a VWF-containing product over screening through study completion (6 months)
  VWF-containing products: Active substances: VWF concentrates, VWF/FVIII concentrates, Cryoprecipitate VWF-containing products licensed in each participating country
Arm/Group | Patients Undergoing On-demand Treatment With a VWF-containing Product
Number analyzed (Participants) | 42
Bleeding events per year | 21.19 (19.337)

3. Secondary Outcome: Consumption of the VWF-containing Product
Description: Data on the consumption of the VWF-containing product (VWF/FVIII IU/kg per month per patient) used for routine on-demand treatment
Time Frame: Screening through study completion (6 months)
Population: Four subjects were not treated with VCP, for two subjects the dose administered is unknown for all infusions
Measure: Mean (Standard Deviation); unit: IUs per kg per month per patient
Arm/Group | Patients Undergoing On-demand Treatment With a VWF-containing Product
Number analyzed (Participants) | 50
IUs per kg per month per patient | 77.94 (67.898)

4. Secondary Outcome: Number of Bleeding Episodes (BEs) Based on a 4-point Efficacy Scale
Description: The efficacy assessment of bleeding episodes at the end of a BE was evaluated on a 4 point scale by the patient/legal guardian (together with the Investigator in case of on-site treatment) including the four items 'excellent,' 'good,' moderate,' and 'none.' The assessment was excellent when bleeding was completely stopped within 3 days in case of minor bleed, within 7 days in case of major bleed, and within 10 days in case of gastrointestinal bleed; Good when bleeding was completely stopped, but time and/or dose slightly exceeded expectations ; Moderate when bleeding could be stopped only by significantly exceeding time and/or dose expectations; and None when bleeding could be stopped only by using other VWF-containing products.
Time Frame: Screening through study completion (6 months)
Population: 39 patients who received VWF-containing product in the treatment of BEs
Measure: Number; unit: Number of Bleeding Episodes
Units Other Than Participants: Number of Bleeding Episodes
Arm/Group | Patients Undergoing On-demand Treatment With a VWF-containing Product
Number analyzed (Participants) | 39
Number analyzed (Number of Bleeding Episodes) | 457
Number of Bleeding Episodes
  Excellent | 450
  Good | 6
  Moderate | 1
  None | 0

5. Secondary Outcome: Number of Surgery With Successful/Unsuccessful Efficacy Assessment
Description: Effectiveness of VWF-containing product in surgical prophylaxis based on the proportion of surgeries successfully treated. Overall treatment efficacy will be assessed at the end of the postoperative period by the treating physician using predefined criteria of 'Excellent', 'Good', 'Moderate/Poor' or 'None'.
Time Frame: From start of surgery until end of post-operative period (within 8 days after surgery)
Population: 6 patients had 7 surgeries that were treated with VWF
Measure: Number; unit: Surgeries
Units Other Than Participants: Number of Surgeries
Groups:
- Patients Undergoing Treatment With a VWF-containing Product for a Surgical Procedure: Patients with type 3, type 2 (except 2N), or severe type 1 VWD undergoing routine on-demand treatment with a VWF-containing product over a period of 6 months
  VWF-containing products: Active substances: VWF concentrates, VWF/FVIII concentrates, Cryoprecipitate VWF-containing products licensed in each participating country
Arm/Group | Patients Undergoing Treatment With a VWF-containing Product for a Surgical Procedure
Number analyzed (Participants) | 6
Number analyzed (Number of Surgeries) | 7
Surgeries
  Excellent | 7
  Good | 0
  Moderate | 0
  Poor | 0

6. Secondary Outcome: Quality of Life (QoL) Assessed Using the Patient-Reported Outcomes Measurement Information System (PROMIS-29)
Description: QoL assessment based on the results from the PROMIS-29 survey to monitor and evaluate the physical, mental, and social health in all patients, using a scale of a minimum score of 0 and a maximum score of 10, with higher scores representing a better outcome. The survey covers seven domains from the most relevant areas of self-reported health (depression, anxiety, physical function, pain interference, fatigue, sleep disturbance and ability to participate in social roles and activities) for the majority of people with chronic illness. PROMIS scores have a mean of 50 and standard deviation (SD) of 10 in a referent population. Full details of cut off points for each domain can be found here: https://www.healthmeasures.net/score-and-interpret/interpret-scores/promis/promis-score-cut-points
Time Frame: At screening visit
Measure: Mean (Standard Deviation); unit: T-Scores
Arm/Group | Patients Undergoing On-demand Treatment With a VWF-containing Product
Number analyzed (Participants) | 56
T-Scores
  Physical Function | 47.24 (7.947)
  Anxiety/Fear | 53.57 (9.941)
  Depression/Sadness | 49.96 (9.265)
  Fatigue | 49.77 (11.202)
  Sleep Disturbance | 49.81 (10.373)
  Ability to Participate in Social Roles/Activities | 52.78 (9.817)
  Pain Interference | 53.87 (11.134)

7. Secondary Outcome: Quality of Life (QoL) Assessed Using a 36-Item Short Form Health Survey, Version 2 (SF-36v2)
Description: QoL assessment based on the results from the SF-36v2 questionnaire to measure functional health and well-being in patients ≥16 years. SF-36v2 ranks 8 different domains using a scale standardized with a scoring algorithm to obtain a score ranging from 0 to 100.The eight health domains include physical functioning (PF), role physical (RP), bodily pain (BP), general health problems (GH), vitality (VT), social functioning (SF), role emotional (RE) and general mental health (MH). Higher scores indicate better health status, and a mean score of 50 has been articulated as a normative value for all scales.
Time Frame: At screening visit
Population: 31 patients complete SF-36 questionnaire
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Patients Undergoing Treatment With a VWF-containing Product: Patients with type 3, type 2 (except 2N), or severe type 1 VWD undergoing routine on-demand treatment with a VWF-containing product over a period of 6 months
  VWF-containing products: Active substances: VWF concentrates, VWF/FVIII concentrates, Cryoprecipitate VWF-containing products licensed in each participating country
Arm/Group | Patients Undergoing Treatment With a VWF-containing Product
Number analyzed (Participants) | 31
Units on a scale
  Bodily Pain | 49.87 (27.304)
  General Health | 49.45 (21.857)
  Mental Health | 62.74 (16.923)
  Physical Functioning | 64.03 (24.509)
  Role Emotional | 62.63 (27.035)
  Role Physical | 51.21 (25.435)
  Social Functioning | 64.52 (24.173)
  Vitality | 58.06 (18.128)

8. Secondary Outcome: Quality of Life (QoL) Assessed Using a 10-item Short Form Health Survey (SF-10)
Description: QoL assessment based on the results from a SF-10 parent-completed questionnaire for patients ≥5.5 and <16 years of age, in order to score physical and psychosocial health. SF-10 uses norm-based scoring where scales have a standardized mean value of 50 and standard deviation of 10.
Time Frame: At screening
Population: 25 subjects completed SF-10 questionnaire
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Patients Undergoing On-demand Treatment With a VWF-containing Product
Number analyzed (Participants) | 25
Units on a scale
  Physical Summary Score | 28.60 (14.961)
  Psychosocial Summary Score | 46.56 (9.428)

9. Secondary Outcome: Joint Health Status Assessed Using Hemophilia Joint Health Score (HJHS)
Description: Joint health status will be assessed using the Hemophilia Joint Health Score (HJHS), which has been specifically validated for the assessment of the clinical outcome in VWD. HJHS evaluates six index joints to produce a score between 0-124. Higher scores indicate worse joint health.
Time Frame: At screening
Population: 37 patients from 42 patients in the PP set completed HJHS
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Patients Undergoing On-demand Treatment With a VWF-containing Product
Number analyzed (Participants) | 37
Units on a scale | 6.76 (14.611)

10. Secondary Outcome: Menstrual Bleeding Assessed Using Pictorial Blood Loss Assessment Chart (PBAC) Score
Description: Bleeding information from each menstrual period while in this study will be collected using the Pictorial Blood Loss Assessment Chart (PBAC). The PBAC will be provided to all female patients of child-bearing potential. The data documented in the PBAC and the investigator-calculated final score will be recorded in the eCRF. The PBAC records pad and tampon use (as either light [1 point], medium [5 points], or heavy [10 points] flow), clots (small [1 point] or large [5 points]), and flooding episodes (1 point each) which can be recorded as many times as necessary any day of the month. The PBAC is scored from 0 (no bleeding) onwards, with a score of >100 defining abnormal coagulation and heavy menstrual bleeding (corresponds to >80ml of blood loss per menstrual cycle).
Time Frame: Screening through study completion (6 months)
Population: All subjects of child bearing potential who experienced menstrual cycle
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Patients Undergoing Treatment With a VWF-containing Product
Number analyzed (Participants) | 15
Units on a scale
  MC01 | 521.7 (790.96)
  MC02: number analyzed (Participants) | 14
  MC02 | 279.2 (219.69)
  MC03: number analyzed (Participants) | 12
  MC03 | 311.0 (261.98)
  MC04: number analyzed (Participants) | 12
  MC04 | 408.8 (471.92)
  MC05: number analyzed (Participants) | 10
  MC05 | 289.9 (267.53)
  MC06: number analyzed (Participants) | 7
  MC06 | 330.4 (327.02)
  MC07: number analyzed (Participants) | 5
  MC07 | 411.6 (314.99)
  MC08: number analyzed (Participants) | 2
  MC08 | 348.5 (102.53)
  MC09: number analyzed (Participants) | 2
  MC09 | 361.5 (400.93)

11. Secondary Outcome: Number of Participants With Adverse Drug Reactions (ADRs) Associated With Use of Wilate
Description: Noxious and unintended reactions arising from the use of Wilate will be monitored throughout the study.
Time Frame: Screening through study completion (6 months)
Population: All participants that were treated with at least one dose of a VWF-containing product
Measure: Count of Participants; unit: Participants
Groups:
- Patients Undergoing Treatment With a VWF-containing Product: Patients with type 3, type 2 (except 2N), or severe type 1 VWD undergoing routine on-demand treatment with a VWF-containing product over a period of 6 months
  VWF-containing products: Active substances: VWF concentrates, VWF/FVIII concentrates, Cryoprecipitate VWF-containing products licensed in each participating country
  Four subjects did not receive a VWF-containing product during the observation period.
Arm/Group | Patients Undergoing Treatment With a VWF-containing Product
Number analyzed (Participants) | 52
Participants | 0

ADVERSE EVENTS:
Time Frame: 6 Months
Arm/Group | Patients Undergoing Treatment With a VWF-containing Product
All-Cause Mortality (participants affected / at risk) | 0/51
Serious Adverse Events (participants affected / at risk) | 0/51
Other Adverse Events (participants affected / at risk) | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-08-05): https://cdn.clinicaltrials.gov/large-docs/99/NCT04053699/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-25): https://cdn.clinicaltrials.gov/large-docs/99/NCT04053699/SAP_001.pdf